CLINICAL TRIAL: NCT02384226
Title: User Testing and Feedback for a Mobile Health Program for Postpartum Women: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1173; UL1TR001082 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes Mellitus; Preeclampsia; Gestational Hypertension; Pre-term Delivery; Delivery of Small for Gestational Age (SGA) Baby
Keywords: mobile application; postpartum; weight loss
MeSH Terms: conditions — Diabetes, Gestational; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Refine content and delivery of the mHealth delivered lifestyle intervention program through iterative testing with small groups of users who provide feedback through on-line asynchronous focus groups.

DETAILED DESCRIPTION:
Participants are asked to:

* Use mobile app for 4 weeks
* Receive support from the lifestyle coach
* Provide weekly and ongoing feedback via an online asynchronous user group platform on usability, navigability, acceptability, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Body Mass Index (BMI): 25 - 45 kg/m2
* Positive history of one or more of the following complications in most recent singleton pregnancy:

  1. Gestational diabetes mellitus
  2. Preeclampsia (high blood pressure and proteinuria diagnosed after 20 weeks gestation)
  3. Gestational hypertension (new hypertension diagnosed after 20 weeks without proteinuria)
  4. Pre-term delivery (32-37 weeks)
  5. Small for gestational age (<10th percentile for gestational age)
* Able to communicate in English
* Access to and be willing to use a wi-fi enabled iPhone or iPod
* Access to a computer with internet access
* Capable of providing informed consent
* Between 4 weeks and 24 weeks after delivery

Exclusion Criteria:

* Personal history of Type 1 or 2 diabetes
* Personal history of breast cancer or any other type of cancer other than a basal cell skin cancer;
* Personal history of major chronic illness including cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication), kidney disease, liver disease, venous or arterial thromboembolic disease, adrenal insufficiency, depression requiring hospitalization within the past 6 months, or non-pregnancy related illness requiring overnight hospitalization in the past 6 months;
* Underlying disease/treatment that might interfere with participation in/completion of the study (e.g. significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be identified via the Perinatal Clinical & Translational Research Center (CTRC) at the University of Colorado at Anschutz Medical Campus.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Usability of the Application | 4 weeks
  Usability is defined via Young's Mobile Phone Usability Questionnaire (MPUQ) as how easy the app is to use and how easy it is to learn. The investigators will assess components of usability including: 1) learnability (how easy is it to accomplish basic tasks the first time the app is used?); 2) efficiency (once users can use the app, how quickly can they perform tasks?); 3) memorability (if a user returns to an app after not using it for some time, how easy is it to re-establish proficiency?); 4) errors (how many, how severe, how easy to recover?); and 5) satisfaction (how pleasant is it to use the app?).
Engagement with the Application | 4 weeks
  The quantitative assessment of the daily use of the mobile application, including the response to prompts, interactions with lifestyle coach, points earned, and tracking of weight, diet, and physical activity.

SECONDARY OUTCOMES:
Navigability of the Application | 4 weeks
  Navigability is defined via Young's Mobile Phone Usability Questionnaire (MPUQ) as whether people can easily and quickly find what they need. The investigators will assess components of navigability including: 1) Is it relatively easy to move from one part of a task to another? 2) Are the operations of this application (app) simple and uncomplicated? 3) Does the app enable the quick, effective, and economical performance of tasks? 4) Is it easy to access the information that you need? 5) Does the app have all the functions and capabilities you expect it to have? 6) Is it easy to navigate between menus and content?
Acceptability of the Application | 4 weeks
  Acceptability is defined whether the intended audience finds the content accessible-meaning that it is written in a way that is easily understood and resonant for this population of postpartum women.

CONTACTS AND LOCATIONS:
Overall Officials: Jacinda M Nicklas, MD, MPH, MA, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicklas JM, Leiferman JA, Lockhart S, Daly KM, Bull SS, Barbour LA. Development and Modification of a Mobile Health Program to Promote Postpartum Weight Loss in Women at Elevated Risk for Cardiometabolic Disease: Single-Arm Pilot Study. JMIR Form Res. 2020 Apr 9;4(4):e16151. doi: 10.2196/16151. PMID 32271149